CLINICAL TRIAL: NCT02826538
Title: Evaluation Der Intraoperativen Umsetzung Von 3D Geplanten Osteosynthesen Mit Patientenspezifischen Zielvorrichtungen Durch Eine Quantitative Postoperative Erfolgskontrolle
Brief Title: 3D Geplante Osteosynthesen Mit Patientenspezifischen Zielvorrichtungen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties recruiting participants
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D-Osteosynthese-Ziel
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Fracture of Humerus; Fracture of Ulna Radius; Fracture of Clavicle; Fracture of Hand; Fracture of Pelvis; Fracture of Femur; Fracture of Tibia Fibula; Fracture of Skull
MeSH Terms: conditions — Humeral Fractures; Hip Fractures; Femoral Fractures; Skull Fractures | interventions — Fracture Fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient specific guides (Experimental): fracture fixation with 3D planning and use of patient-specific instruments
  Interventions: Device: fracture fixation with patient specific guides
- standard procedure (Active Comparator): standard procedure of fracture Fixation without 3D planning and without use of patient-specific instruments
  Interventions: Device: standard procedure of fracture fixation

INTERVENTIONS:
Device: fracture fixation with patient specific guides — Using the preoperative computed tomography scan, a 3D planning of the fracture Fixation is made and patient-specific guides for fracure fixation are produced using a 3D Printer. These Patient-specific guides are used for fracture fixation
  Other Names: MyOsteotomy
  Arms: patient specific guides
Device: standard procedure of fracture fixation — the standard procedure of fracure fixation for each fracture localisation is used as a standard of reference
  Arms: standard procedure

SUMMARY:
Goal of this study is to evaluate the accuracy of 3D computer-planned fracture fixation with patient-specific instruments for clavicle, upper extremity, lower extremity and pelvis fractures compared with the standard procedure of fracture fixation.

DETAILED DESCRIPTION:
The research hypothesis is: The medical product permits the fracture fixation of clavicle, upper extremity, lower extremity and pelvis fractures to be more accurate compared with standard procedures of fracture fixation. Accuracy is evaluated by calculating translation and rotation comparing the postoperative 3D model versus the preoperative 3D plan.

Secondary outcome is an assessment of the surgical outcome using validated outcome instruments for each fractured body part like "Patient related wrist Evaluation" (PRWE) scores for distal radial fractures, as well as evaluation of range of motion.

ELIGIBILITY:
Inclusion Criteria:

* fracture of clavicle, upper extremity, lower extremity or pelvis,tibia, fibula,Femur, with indication for fracture Fixation
* clinical indication for a computed tomography of the fractured bone
* >18 years of Age
* Patient is able to give informed consent

Exclusion Criteria:

* pregnancy or nursing women
* non-compliance of the patient to follow the clinical study protocol, drug abuse or alcohol abuse
* participation in a different clinical Trial within the last 30 days before inclusion or during the study
* allergy to Polyamid PA 2200
* no available technique for fracture Fixation which could be performed, in case of applying the medical device is not possible.
* Applying the medical device is not possible, because of technical or anatomical reasons.
* other clinical significant accompanying symptoms (tumor, infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
3D difference between preoperative plan and surgery | 12 months
  For each surgery the discrepancy of the postoperative result compared to the preoperative planning is calculated by measuring all 6 degrees of freedom (3xrotation, 3xtranslation). The discrepancy between a simulated perfect postoperative result and the actual postoperative result is assessed in degree (rotation) and millimeters (translation). These measures are used to compare the outcome of the two different study Groups.

SECONDARY OUTCOMES:
surgical outcome assesed by validated outcome instruments | 12 months
  The surgical outcome is assessed by using specific validated outcome instruments for each fracture localisation, for example PRWE-score for wrist fractures.
range of motion | 12 months
  range of Motion is postoperatively assessed and compared between interventional and control group

CONTACTS AND LOCATIONS:
Overall Officials: Phillipp Furnstahl, PhD, Principal Investigator — Balgrist University Hospital; Philipp Furnstahl, PhD, Study Director — Balgrist University Hospital
Locations (2):
- Switzerland (2):
  - Universital Hospital Zurich, Zurich
  - University Hospital Balgrist, Zurich

IPD SHARING:
Plan to Share IPD: Undecided